CLINICAL TRIAL: NCT03736564
Title: 68Ga-DOTATATE PET for Localization of Phosphaturic Mesenchymal Tumors in Patients With Tumor Induced Osteomalacia
Brief Title: Ga-DOTATATE PET for Phosphaturic Mesenchymal Tumors in Patients With Tumor Induced Osteomalacia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-008120; NCI-2023-00775 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-10-30; First posted 2018-11-09 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Osteomalacia
Keywords: FGF 23; oncogenic; tumor induced
MeSH Terms: conditions — Osteomalacia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- 68Ga-DOTATATE PET/CT (Experimental): Subjects will undergo imaging by 68Ga-DOTATATE PET/CT
  Interventions: Combination Product: 68Ga-DOTATATE PET/CT

INTERVENTIONS:
Combination Product: 68Ga-DOTATATE PET/CT — Gallium-68 Dotatate, a radioactive imaging agent, is injected into a vein. Subjects will rest for approximately 50 minutes, after which approximately a 30 minute image of subjects body will be completed via PET/CT scan.

SUMMARY:
The researchers are trying to evaluate a newer imaging technique (Ga-DOTATATE PET/CT) to see if it is more sensitive to localize the source of the hormone, which has caused the low phosphate levels.

DETAILED DESCRIPTION:
Subjects will be contacted (phone script attached) to inform them of the study and the imaging modality. The first 10 patients that agree to participate in the study will be asked to present to the Mayo Clinic where they can provide a written consent and perform the imaging study.

Enrolled subjects will be evaluated in the clinical practice prior to having 68Ga-DOTATATE PET/CT imaging performed. The treating endocrinologist will be informed of the imaging results and will review the results with the subject using a follow-up visit or phone call; when a tumor is localized, the endocrinologist will discuss appropriate management options.

Subjects will be follow for one year post 68Ga-DOTATATE PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years of age or older) seen at Mayo Clinic, Rochester for FGF23 mediated osteomalacia between 1/1/2000 and 1/30/2018 who provide informed consent to participate in the study.

Exclusion Criteria:

* Pregnant
* Prisoners
* Subjects diagnosed with heritable hypophosphatemic rickets/osteomalacia
* Subjects who do not consent for the study or withdraw consent during the duration of the study.
* Subjects in whom tumor localization and successful resection has already occurred.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Drake, MD, Principal Investigator — Mayo Clinic; Stephen M Broski, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 68Ga-DOTATATE PET/CT
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 68Ga-DOTATATE PET/CT
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Positive Localization of Phosphaturic Mesenchymal Tumors (PMTs)
Description: 68Ga-DOTATATE PET maximum intensity projection images will be analyzed to evaluate for the localization of phosphaturic mesenchymal tumors (PMTs).
Time Frame: One year
Measure: Count of Participants; unit: Participants
Arm/Group | 68Ga-DOTATATE PET/CT
Number analyzed (Participants) | 18
Participants | 15

ADVERSE EVENTS:
Time Frame: Participants were monitored from administration of the radioactive imaging agent until approximately 30 minutes after PET/CT scan, for a total of approximately 2 hours.
Arm/Group | 68Ga-DOTATATE PET/CT
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT03736564/Prot_SAP_002.pdf
  • Informed Consent Form (2022-11-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT03736564/ICF_001.pdf